CLINICAL TRIAL: NCT00536471
Title: Duloxetine Versus Placebo in Patients With Major Depressive Disorder (MDD): Assessment of Energy and Vitality in MDD
Brief Title: A Study Comparing Duloxetine and Placebo in Assessing Energy and Vitality in Major Depressive Disorder (MDD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11669; F1J-US-HMFS
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): duloxetine 60 milligrams (mg) every day (QD), by mouth (PO) for 3 months, after which may be increased to duloxetine 120 mg QD, PO for 6 months
  Interventions: Drug: Duloxetine hydrochloride
- B (Placebo Comparator): placebo every day (QD), by mouth (PO) for up to 9 months, may be increased to duloxetine 60 mg QD, PO during the first 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine hydrochloride
  Other Names: LY248686; Cymbalta
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
Study F1J-US-HMFS comprises two identical multicenter, 9-month, randomized, placebo-controlled, double-blind, trials (HMFSa and HMFSb). The purpose of this study is to compare the efficacy and safety of Duloxetine 60 milligrams (mg) once daily to placebo on depression in patients aged 18-65. Data from the two trials will be reported in both individual and pooled analyses. Pooling the two studies will allow for increased power to detect differences between duloxetine and placebo on secondary and exploratory objectives. Only one data lock is planned for this study, when all patients have completed all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients
* Aged 18-65 who meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnostic criteria for Major Depressive Disorder (MDD)
* Have a Montgomery-Asberg Depression Rating Scale (MADRS) total score of at least 22 at visits 1 and 2
* Have a Clinical Global Impressions of Severity Scale (CGI-S) score of at least 4 at visits 1 and 2
* Have a degree of understanding such that the patient can provide informed consent, complete protocol required assessments and communicate intelligibly with the investigator and study coordinator.

Exclusion Criteria:

* Patients judged clinically to be at serious suicidal risk in the opinion of the investigator
* Patients who have any prior history of bipolar disorder, psychosis, or schizophrenia
* Patients who have any current (within the past six months) DSM-IV-TR primary Axis I disorder other than MDD
* Patients with uncontrolled narrow-angle glaucoma
* Patients who have a serious medical illness that is in the opinion of the investigator not stabilized or is likely to require intervention, hospitalization, or use of an excluded medication during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (47):
- United States (43):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New London, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edwardsville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naperville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., City of Saint Peters, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Allis, Wisconsin
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arecibo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- [Derived] Harada E, Kato M, Fujikoshi S, Wohlreich MM, Berggren L, Tokuoka H. Changes in energy during treatment of depression: an analysis of duloxetine in double-blind placebo-controlled trials. Int J Clin Pract. 2015 Oct;69(10):1139-48. doi: 10.1111/ijcp.12658. Epub 2015 May 16. PMID 25980552
- [Derived] Dodd S, Berk M, Kelin K, Zhang Q, Eriksson E, Deberdt W, Craig Nelson J. Application of the Gradient Boosted method in randomised clinical trials: Participant variables that contribute to depression treatment efficacy of duloxetine, SSRIs or placebo. J Affect Disord. 2014 Oct;168:284-93. doi: 10.1016/j.jad.2014.05.014. Epub 2014 Jun 4. PMID 25080392
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study HMFS comprises two identical trials (identified as Group A and Group B). Study Period I was a screening period. Study Period II was a 9-month double-blind treatment period. Study Period III was an optional double-blind 2-week discontinuation/taper period.
Groups:
- Group A - Duloxetine; Group B - Duloxetine: duloxetine 60 mg every day (QD), by mouth (PO) for 3 months, after which may be increased to duloxetine 120 mg QD, PO for 6 months
- Group A - Placebo; Group B - Placebo: placebo every day (QD), by mouth (PO) for up to 9 months, may be increased to duloxetine 60 mg QD, PO during the first 3 months as part of a rescue plan with pre-defined criteria (Patients meeting criteria will automatically be assigned to duloxetine 60 mg QD).
Period: Overall Study
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Started | 257 | 127 | 261 | 131
Completed | 101 | 43 | 122 | 57
Not Completed | 156 | 84 | 139 | 74
Not completed — Lost to Follow-up | 48 | 23 | 48 | 22
Not completed — Adverse Event | 32 | 16 | 28 | 13
Not completed — Withdrawal by Subject | 40 | 24 | 43 | 21
Not completed — Lack of Efficacy | 17 | 18 | 11 | 9
Not completed — Protocol Violation | 8 | 1 | 2 | 3
Not completed — Physician Decision | 11 | 1 | 3 | 2
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Sponsor Decision | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo | Total
Number analyzed (Participants) | 257 | 127 | 261 | 131 | 776
Age Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.2) | 43.7 (12.5) | 44.7 (12.2) | 43.9 (11.9) | 43.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 78 | 169 | 87 | 489
  Male | 102 | 49 | 92 | 44 | 287
Region of Enrollment [Number; unit: participants]
  United States | 249 | 123 | 222 | 110 | 704
  Puerto Rico | 8 | 4 | 39 | 21 | 72
History - Atypical Depression [Number; unit: participants]
  Yes | 7 | 5 | 19 | 7 | 38
  No | 250 | 122 | 242 | 124 | 738
History - Melancholic Depression [Number; unit: participants]
  Yes | 134 | 71 | 147 | 71 | 423
  No | 123 | 56 | 114 | 60 | 353
History - Seasonal Pattern in Major Depressive Disorder (MDD) if ≥3 Previous MDD Episodes [Number; unit: participants]
  Yes | 3 | 3 | 9 | 4 | 19
  No | 220 | 105 | 232 | 112 | 669
  Missing Response | 34 | 19 | 20 | 15 | 88
Race/Ethnicity [Number; unit: participants]
  African | 63 | 36 | 30 | 16 | 145
  Caucasian | 160 | 73 | 172 | 81 | 486
  Hispanic | 29 | 11 | 55 | 30 | 125
  East Asian | 3 | 5 | 3 | 1 | 12
  West Asian (Indian sub-continent) | 2 | 2 | 1 | 2 | 7
  Native American | 0 | 0 | 0 | 1 | 1
Body Height [Mean (Standard Deviation); unit: centimeters] | 168.1 (10.1) | 168.5 (9.2) | 169.0 (9.7) | 168.8 (9.4) | 168.6 (9.7)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 88.8 (23.7) | 84.9 (22.5) | 88.6 (26.6) | 86.4 (23.5) | 87.7 (24.5)
Evaluation - Brief Profile of Mood States (BPOMS) [Mean (Standard Deviation); unit: units on a scale] — The 30-item BPOMS measures mood states and has 6 factors: tension-anxiety, depression-dejection, anxiety-hostility, fatigue, confusion, and vigor. Item scores: 0 (not at all) to 4 (extremely). Each factor scores range from 0 to 20. The Total score is sum of all factor scores minus the factor score for vigor (Total=Ten+Dep+Ang+Fat+Con-Vig).
  units on a scale
    Total Score | 49.0 (19.2) | 47.5 (18.7) | 51.8 (19.3) | 51.8 (18.7) | 50.2 (19.1)
    Tension-Anxiety Score | 9.5 (4.6) | 9.2 (4.6) | 10.0 (5.0) | 10.4 (4.6) | 9.8 (4.7)
    Depression-Dejection Score | 11.8 (4.8) | 11.5 (4.8) | 12.3 (4.6) | 12.0 (4.2) | 12.0 (4.7)
    Anger-Hostility Score | 8.9 (5.4) | 9.0 (5.4) | 9.5 (5.1) | 9.5 (5.4) | 9.2 (5.3)
    Vigor-Activity Score | 3.4 (3.1) | 3.9 (3.1) | 3.6 (3.5) | 3.4 (3.0) | 3.5 (3.2)
    Fatigue-Inertia Score | 12.8 (4.6) | 12.3 (4.8) | 13.5 (4.7) | 13.2 (4.5) | 13.0 (4.7)
    Confusion-Bewilderment Score | 9.7 (4.0) | 9.6 (3.9) | 9.8 (4.1) | 10.1 (3.8) | 9.8 (4.0)
Evaluation - 16-Item Quick Inventory of Depressive Symptomatology (QIDS16) Total Score [Mean (Standard Deviation); unit: units on a scale] — A 16-item patient-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity.
  units on a scale | 14.7 (4.1) | 13.7 (4.4) | 15.0 (4.4) | 14.7 (3.8) | 14.6 (4.2)
Evaluation - 17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 22.9 (4.3) | 22.8 (3.7) | 22.8 (4.5) | 22.9 (4.9) | 22.8 (4.4)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 10:Anxiety (Psychic) [Mean (Standard Deviation); unit: units on a scale] — Measures anxiety on a scale of 0 (no difficulty) to 4 (fears expressed).
  units on a scale | 2.1 (0.8) | 2.1 (0.7) | 2.1 (0.8) | 2.2 (0.8) | 2.1 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 11:Anxiety (Somatic) [Mean (Standard Deviation); unit: units on a scale] — Measures physiological concomitants of anxiety on a scale of 0 (absent) to 4 (incapacitating).
  units on a scale | 1.4 (0.8) | 1.5 (0.8) | 1.6 (0.9) | 1.6 (0.9) | 1.5 (0.9)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 13:Somatic Symptoms/General [Mean (Standard Deviation); unit: units on a scale] — Measures general somatic symptoms on a scale of 0 (none) to 2 (any clear-cut symptoms).
  units on a scale | 1.6 (0.6) | 1.7 (0.5) | 1.7 (0.5) | 1.7 (0.6) | 1.7 (0.5)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 14:Genital Symptoms [Mean (Standard Deviation); unit: units on a scale] — Measures genital symptoms (loss of libido, menstrual disturbances) on a scale of 0 (absent) to 2 (severe).
  units on a scale | 1.3 (0.8) | 1.2 (0.9) | 1.3 (0.8) | 1.1 (0.9) | 1.2 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 15:Hypochondriasis [Mean (Standard Deviation); unit: units on a scale] — Measures hypochondriasis on a scale of 0 (not present) to 4 (hypochondriacal delusions).
  units on a scale | 0.7 (0.8) | 0.7 (0.8) | 1.0 (0.9) | 1.1 (0.9) | 0.9 (0.9)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 16:Loss of Weight [Mean (Standard Deviation); unit: units on a scale] — Measures weight loss since last visit on a scale of 0 (no weight loss) to 2 (definite weight loss caused by present illness).
  units on a scale | 0.3 (0.6) | 0.2 (0.5) | 0.3 (0.6) | 0.4 (0.7) | 0.3 (0.6)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 17:Insight [Mean (Standard Deviation); unit: units on a scale] — Measures insight on a scale of 0 (acknowledges being depressed and ill) to 2 (denies being ill at all).
  units on a scale | 0.2 (0.4) | 0.2 (0.4) | 0.1 (0.2) | 0.0 (0.2) | 0.1 (0.4)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 18A:Diurnal Variation [Mean (Standard Deviation); unit: units on a scale] — Measures whether symptoms are worse in morning or evening on a scale of 0 (no variation), 1 (worse in morning), or 2 (worse in evening).
  units on a scale | 0.8 (0.8) | 0.9 (0.9) | 1.0 (0.9) | 1.0 (0.9) | 0.9 (0.9)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 1:Depressed Mood [Mean (Standard Deviation); unit: units on a scale] — Measures depressed mood on a scale of 0 (absent) to 4 (very depressed).
  units on a scale | 3.0 (0.6) | 2.9 (0.6) | 2.9 (0.6) | 2.9 (0.5) | 2.9 (0.6)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 20:Paranoid Symptoms [Mean (Standard Deviation); unit: units on a scale] — Measures paranoid symptoms on a scale of 0 (none) to 3 (delusions of reference and persecution).
  units on a scale | 0.2 (0.5) | 0.2 (0.5) | 0.2 (0.5) | 0.2 (0.4) | 0.2 (0.5)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 22B:Helplessness [Mean (Standard Deviation); unit: units on a scale] — Measures feelings of helplessness on a scale of 0 (absent) to 4 (severe).
  units on a scale | 1.4 (1.0) | 1.5 (1.0) | 1.5 (1.0) | 1.7 (1.0) | 1.5 (1.0)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 23B:Hopelessness [Mean (Standard Deviation); unit: units on a scale] — Measures feelings of hopelessness on a scale of 0 (absent) to 3 (expresses feelings of discouragement, despair, and/or pessimism about the future which cannot be dispelled).
  units on a scale | 1.3 (0.8) | 1.3 (0.9) | 1.3 (0.8) | 1.3 (0.9) | 1.3 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 24B:Worthlessness [Mean (Standard Deviation); unit: units on a scale] — Measures feelings of worthlessness on a scale of 0 (absent) to 4 (severe).
  units on a scale | 1.5 (1.0) | 1.5 (1.0) | 1.6 (1.1) | 1.6 (1.1) | 1.5 (1.0)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 2:Feelings of Guilt [Mean (Standard Deviation); unit: units on a scale] — Measures feelings of guilt on a scale of 0 (absent) to 4 (very guilty).
  units on a scale | 1.8 (0.7) | 2.0 (0.7) | 1.8 (0.6) | 1.7 (0.8) | 1.8 (0.7)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 3:Suicide [Mean (Standard Deviation); unit: units on a scale] — Measures thoughts of suicide on a scale of 0 (absent) to 4 (attempts suicide).
  units on a scale | 0.6 (0.7) | 0.7 (0.7) | 0.6 (0.8) | 0.6 (0.8) | 0.6 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 4:Insomnia Early [Mean (Standard Deviation); unit: units on a scale] — Measures early insomnia on a scale of 0 (no difficulty falling asleep) to 2 (complains of nightly difficulty falling asleep).
  units on a scale | 1.5 (0.8) | 1.4 (0.8) | 1.4 (0.8) | 1.4 (0.8) | 1.4 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 5:Insomnia Middle [Mean (Standard Deviation); unit: units on a scale] — Measures middle insomnia on a scale of 0 (no difficulty) to 2 (waking during the night).
  units on a scale | 1.5 (0.7) | 1.5 (0.6) | 1.4 (0.8) | 1.5 (0.7) | 1.5 (0.7)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 6:Insomnia Late [Mean (Standard Deviation); unit: units on a scale] — Measures late insomnia on a scale of 0 (no difficulty) to 2 (unable to fall asleep again if gets out of bed).
  units on a scale | 1.2 (0.8) | 1.3 (0.8) | 1.1 (0.8) | 1.1 (0.8) | 1.2 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 7:Work and Activities [Mean (Standard Deviation); unit: units on a scale] — Item 7 of the HAMD-24 assesses loss of interest or pleasure in work and activities and is an essential symptom in MDD. Scores range from 0 (no difficulty/no loss) to 4 (difficulty/loss).
  units on a scale | 2.9 (0.5) | 2.8 (0.6) | 2.8 (0.5) | 2.8 (0.5) | 2.8 (0.5)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 8:Retardation [Mean (Standard Deviation); unit: units on a scale] — Measures slowness of thought and speech; impaired ability to concentrate; decreased motor activity on a scale of 0 (normal speech and thought) to 4 (complete stupor).
  units on a scale | 1.1 (0.7) | 1.0 (0.7) | 1.1 (0.8) | 1.1 (0.9) | 1.1 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) - Item 9:Agitation [Mean (Standard Deviation); unit: units on a scale] — Measures agitation on a scale of 0 (none) to 4 (hand-wringing, nail-biting).
  units on a scale | 0.9 (0.9) | 0.9 (0.8) | 0.9 (0.9) | 1.0 (0.9) | 0.9 (0.9)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Anxiety/Somatization Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Anxiety/Somatization subscale (items 10-13, 15, 17) evaluates severity of psychic and somatic manifistations of anxiety as well as agitation. Total subscale scores range from 0 (normal) to 18 (severe).
  units on a scale | 6.8 (2.1) | 6.9 (1.9) | 7.1 (2.3) | 7.3 (2.4) | 7.0 (2.2)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Bech Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Bech subscale (Items 1,2,7,8,10,13) evaluates "core" symptoms of Major Depressive Disorder (MDD). Total subscale scores range from 0 (normal) to 22 (severe).
  units on a scale | 12.6 (2.0) | 12.5 (1.7) | 12.4 (1.9) | 12.3 (2.2) | 12.5 (2.0)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Maier Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Maier subscale (Items 1,2,7,8,9,10) represents the "core" symptoms of depression. Total subscale scores range from 0 (normal) to 24 (severe).
  units on a scale | 11.8 (2.2) | 11.7 (1.9) | 11.6 (2.2) | 11.6 (2.4) | 11.7 (2.2)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Retardation Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Retardation subscale (Items 1,7,8,14) evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation. Total subscale scores range from 0 (normal) to 14 (severe).
  units on a scale | 8.2 (1.6) | 8.0 (1.6) | 8.0 (1.6) | 7.9 (1.6) | 8.1 (1.6)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Sleep Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Sleep subscale (Items 4,5,6) evaluates initial, middle, and late insomnia. Total subscale scores range from 0 (no difficulty) to 6 (difficulty).
  units on a scale | 4.2 (1.6) | 4.3 (1.5) | 3.9 (1.7) | 4.0 (1.5) | 4.1 (1.6)
Evaluation - 24-Item Hamilton Depression Rating Scale (HAMD-24) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 24-item HAMD measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76.
  units on a scale | 28.6 (6.0) | 28.6 (5.5) | 28.7 (6.2) | 29.0 (6.7) | 28.7 (6.1)
Evaluation - 24-Item Hamilton Depression Rating Scale - Item 12:Somatic Symptoms/Gastrointestinal [Mean (Standard Deviation); unit: units on a scale] — Measures gastrointestical somatic symptoms on a scale of 0 (none) to 2 (difficulty eating, requires medication for symptoms).
  units on a scale | 0.7 (0.7) | 0.6 (0.7) | 0.6 (0.7) | 0.7 (0.7) | 0.7 (0.7)
Evaluation - 24-Item Hamilton Depression Rating Scale - Item 18B:Diurnal Variation-Severity [Mean (Standard Deviation); unit: units on a scale] — Measures the severity of the diurnal variation on a scale of 0 (none) to 2 (severe).
  units on a scale | 0.8 (0.8) | 0.9 (0.9) | 0.9 (0.8) | 1.0 (0.9) | 0.9 (0.8)
Evaluation - 24-Item Hamilton Depression Rating Scale - Item 19: Depersonalization and Derealization [Mean (Standard Deviation); unit: units on a scale] — Measures feelings of unreality on a scale of 0 (absent) to 4 (incapacitating).
  units on a scale | 0.2 (0.6) | 0.3 (0.6) | 0.2 (0.5) | 0.2 (0.5) | 0.2 (0.6)
Evaluation - 24-Item Hamilton Depression Rating Scale - Item 21:Obsessional and Compulsive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Measures obsessional and compulsive symptoms on a scale of 0 (absent) to 2 (severe).
  units on a scale | 0.1 (0.4) | 0.1 (0.4) | 0.1 (0.4) | 0.1 (0.4) | 0.1 (0.4)
Evaluation - Clinical Global Impressions of Severity Scale (CGI-S) Score [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
  units on a scale | 4.6 (0.6) | 4.5 (0.6) | 4.7 (0.7) | 4.7 (0.7) | 4.6 (0.7)
Evaluation - Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire [Mean (Standard Deviation); unit: units on a scale] — A 7-item patitent-rated questionnaire pertaining to a patient's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each of the 7 questions is scored on a 6-point scale ranging fom 1 (greater than normal) to 6 (totally absent). Total score ranges from 7 to 42.
  units on a scale | 28.4 (6.0) | 26.8 (6.1) | 28.6 (6.1) | 28.6 (5.4) | 28.2 (6.0)
Evaluation - Pain Numerical Rating Scale (NRS) Score Item 1 [Mean (Standard Deviation); unit: units on a scale] — Item 1=Average musculoskeletal pain severity. Participants are asked to rate their average pain over the last week as measured by an 11-point Likert scale. A score of 0 reflects "no pain" and a score of 10 reflects "worst possible pain".
  units on a scale | 4.3 (2.8) | 4.1 (2.7) | 4.5 (3.1) | 4.5 (2.8) | 4.4 (2.9)
Evaluation - Pain Numerical Rating Scale (NRS) Score Item 7 [Mean (Standard Deviation); unit: units on a scale] — Item 7=How much they have been bothered by pain over the last week, as measured by an 11-point Likert scale. A score of 0 reflects "not bothered at all" and a score of 10 reflects "extremely bothered".
  units on a scale | 4.7 (3.0) | 4.5 (3.1) | 4.7 (3.2) | 4.9 (3.2) | 4.7 (3.1)
Evaluation - Sheehan Disability Scale (SDS) Item 1 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the patient and Item 1 is used to assess the effect of the patient's symptoms on their work/school schedule. Scores range from 0 to 10 with higher values indicating greater disruption in the patient's work/school life.
  units on a scale | 5.5 (2.8) | 5.4 (2.7) | 5.6 (2.7) | 5.3 (2.8) | 5.5 (2.7)
Evaluation - Sheehan Disability Scale (SDS) Item 2 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the patient and Item 2 is used to assess the effect of the patient's symptoms on their social life/leisure acitivities. Scores range from 0 to 10 with higher values indicating greater disruption in the patient's social life.
  units on a scale | 6.6 (2.4) | 6.2 (2.8) | 6.4 (2.8) | 5.9 (2.5) | 6.3 (2.6)
Evaluation - Sheehan Disability Scale (SDS) Item 3 [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the patient and Item 3 is used to assess the effect of the patient's symptoms on their family life/home responsibilities. Scores range from 0 to 10 with higher values indicating greater disruption in the patient's family life/home responsibilities.
  units on a scale | 6.5 (2.5) | 6.0 (2.6) | 6.2 (2.6) | 6.0 (2.5) | 6.2 (2.6)
Evaluation - Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life.
  units on a scale | 19.0 (6.5) | 17.8 (7.3) | 18.4 (7.1) | 17.5 (7.0) | 18.3 (6.9)
Evaluation - Social Adaptation Self-Evaluation Scale (SASS) Total [Mean (Standard Deviation); unit: units on a scale] — A 21-item self-rated scale that evaluates patient social motivation and behavior in depression. Each of the 21 items is scored from 0 (minimal social adjustment) to 3 (maximal social adjustment). Total score ranges from 0 to 60.
  units on a scale | 27.2 (7.3) | 29.1 (8.4) | 27.6 (8.2) | 29.3 (8.2) | 28.0 (8.0)
History - Age at First Episode [Mean (Standard Deviation); unit: years] | 30.0 (13.2) | 31.2 (13.7) | 30.7 (13.6) | 30.0 (12.6) | 30.4 (13.3)
History - How Long was Last Major Depressive Disorder (MDD) Episode [Mean (Standard Deviation); unit: weeks] | 4.7 (6.3) | 5.0 (7.4) | 5.2 (6.9) | 6.5 (14.5) | 5.2 (8.6)
History - Interval Between Start of Current and Remission of Last MDD Episode [Mean (Standard Deviation); unit: weeks] | 13.2 (20.1) | 12.5 (24.3) | 13.1 (22.1) | 13.1 (22.2) | 13.0 (21.8)
History - Number of Previous Episodes [Mean (Standard Deviation); unit: number of previous episodes] | 4.0 (4.8) | 3.8 (4.3) | 4.9 (5.4) | 5.2 (5.4) | 4.5 (5.1)
History - Time Since First Episode Date [Mean (Standard Deviation); unit: years] | 12.3 (11.6) | 12.5 (11.6) | 14.0 (11.5) | 14.0 (12.0) | 13.2 (11.7)
History - Time Since Most Recent Episode [Mean (Standard Deviation); unit: weeks] | 44.0 (60.2) | 48.8 (69.5) | 51.4 (103.3) | 59.2 (111.2) | 49.8 (87.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 8 Weeks in 24-Item Hamilton Depression Rating Scale (HAMD-24) Item 7 (Work and Activities)
Description: Item 7 of the HAMD-24 assesses loss of interest or pleasure in work and activities and is an essential symptom in MDD. Scores range from 0 (no difficulty/no loss) to 4 (difficulty/loss).
Time Frame: baseline, 8 weeks
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 214 | 102 | 220 | 110
units on a scale | -1.32 (0.07) | -1.07 (0.11) | -1.37 (0.07) | -0.93 (0.09)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis — Repeated Measures Analysis for Group A change from baseline to 8 week endpoint; Model=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Repeated Measures Analysis for Group B change from baseline to 8 week endpoint; Model=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit

2. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in the 17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score and HAMD-24 Subscales (8 Week Endpoint for Maier Subscale)
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe). Please see baseline demographics for subscale total scores.
Time Frame: Baseline, 8 weeks, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 214 | 102 | 220 | 110
units on a scale
  Total Score 12 Week Change (n=194,n=59,n=195,n=64) | -12.64 (0.50) | -10.33 (0.79) | -12.11 (0.47) | -8.48 (0.75)
  Maier 8 Week Change (n=214,n=102,n=220,n=110) | -6.11 (0.27) | -4.69 (0.38) | -6.13 (0.24) | -4.45 (0.33)
  Anxiety 12 Week Change (n=194,n=59,n=195,n=64) | -3.52 (0.16) | -3.12 (0.27) | -3.52 (0.17) | -2.44 (0.27)
  Bech 12 Week Change (n=194,n=59,n=195,n=64) | -7.38 (0.29) | -6.17 (0.47) | -6.98 (0.27) | -4.70 (0.43)
  Retardation 12 Week Change (n=194,n=59,n=195,n=64) | -4.72 (0.19) | -4.06 (0.32) | -4.49 (0.19) | -3.05 (0.31)
  Sleep 12 Week Change (n=194,n=59,n=195,n=64) | -2.08 (0.13) | -1.72 (0.22) | -1.91 (0.12) | -1.48 (0.20)
  Total Score 9 Month Change (n=29,n=9,n=33,n=10) | -14.38 (1.02) | -13.38 (1.86) | -9.56 (1.26) | -5.92 (2.32)
  Anxiety 9 Month Change (n=29,n=9,n=33,n=10) | -4.09 (0.30) | -3.88 (0.56) | -3.44 (0.35) | -2.77 (0.65)
  Bech 9 Month Change (n=29,n=9,n=33,n=10) | -8.56 (0.58) | -8.02 (1.04) | -5.80 (0.70) | -4.35 (1.30)
  Retardation 9 Month Change (n=29,n=9,n=33,n=10) | -5.35 (0.40) | -5.83 (0.72) | -3.68 (0.44) | -2.52 (0.81)
  Sleep 9 Month Change (n=29,n=9,n=33,n=10) | -2.77 (0.23) | -2.56 (0.40) | -2.55 (0.26) | -1.95 (0.48)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — P-value for Total Score 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis — P-value for Maier 8 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.202, Mixed Models Analysis — P-value for Anxiety/Somatization 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — P-value for Bech 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 7]
Statistical Analysis 9: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis — P-value for Retardation 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 10: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 9]
Statistical Analysis 11: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.149, Mixed Models Analysis — P-value for Sleep 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 12: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 11]
Statistical Analysis 13: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.629, Mixed Models Analysis — P-value for Total Score 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 14: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.194, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 13]
Statistical Analysis 15: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.525, Mixed Models Analysis — P-value for Maier 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 16: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.595, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 15]
Statistical Analysis 17: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.736, Mixed Models Analysis — P-value for Anxiety/Somatization 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 18: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 17]
Statistical Analysis 19: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.660, Mixed Models Analysis — P-value for Bech 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 20: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.334, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 19]
Statistical Analysis 21: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.568, Mixed Models Analysis — P-value for Retardation 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 22: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.216, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 21]
Statistical Analysis 23: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.646, Mixed Models Analysis — P-value for Sleep 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit
Statistical Analysis 24: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.275, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 23]

3. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in the HAMD-24 Total Score
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 193 | 57 | 194 | 64
units on a scale
  12 Week Change | -16.24 (0.62) | -13.24 (1.01) | -15.60 (0.61) | -10.94 (0.96)
  9 Month Change (n=29, n=8, n=32, n=10) | -17.05 (1.15) | -15.22 (2.14) | -13.49 (1.45) | -9.12 (2.64)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — P-value for 12 Week Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.449, Mixed Models Analysis — P-value for 9 Month Change. Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.167, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 3]

4. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in the HAMD-24 Item 1:Depressed Mood
Description: Measures depressed mood on a scale of 0 (absent) to 4 (very depressed).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -1.86 (0.07) | -1.52 (0.12) | -1.78 (0.07) | -1.15 (0.12)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.44 (0.20) | -1.26 (0.34) | -1.98 (0.19) | -1.65 (0.35)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for 12 Week Change (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.653, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for 9 Month Change (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.417, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

5. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 2:Feelings of Guilt
Description: Measures feelings of guilt on a scale of 0 (absent) to 4 (very guilty).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -1.19 (0.06) | -1.06 (0.09) | -1.15 (0.05) | -0.89 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.32 (0.10) | -1.21 (0.17) | -1.37 (0.06) | -1.16 (0.13)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for 12 Week Change(Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

6. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 3:Suicide
Description: Measures thoughts of suicide on a scale of 0 (absent) to 4 (attempts suicide).
Time Frame: Baseline, 12 weeks, 9 Months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.46 (0.04) | -0.30 (0.06) | -0.40 (0.04) | -0.29 (0.06)
  9 Month Change (n=29, n= 9, n=33, n=10) | -1.32 (0.10) | -1.21 (0.17) | -1.37 (0.06) | -1.16 (0.13)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.100, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

7. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 4:Insomnia Early
Description: Measures early insomnia on a scale of 0 (no difficulty falling asleep) to 2 (complains of nightly difficulty falling asleep).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.72 (0.06) | -0.61 (0.10) | -0.68 (0.06) | -0.46 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.85 (0.13) | -0.77 (0.23) | -0.71 (0.13) | -0.86 (0.24)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.332, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.775, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.588, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

8. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 5:Insomnia Middle
Description: Measures middle insomnia on a scale of 0 (no difficulty) to 2 (waking during the night).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.69 (0.05) | -0.74 (0.09) | -0.66 (0.06) | -0.59 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.99 (0.11) | -0.92 (0.19) | -0.99 (0.09) | -0.67 (0.16)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.624, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.473, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.787, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

9. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 6:Insomnia Late
Description: Measures late insomnia on a scale of 0 (no difficulty) to 2 (unable to fall asleep again if gets out of bed).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.66 (0.05) | -0.49 (0.09) | -0.57 (0.05) | -0.45 (0.08)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.94 (0.05) | -0.87 (0.08) | -0.78 (0.10) | -0.52 (0.19)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.223, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.473, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.233, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

10. Secondary Outcome: Change From Baseline to 9 Month Endpoint in HAMD-24 - Item 7:Work and Activities
Description: as for outcome 1
Time Frame: Baseline, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 29 | 9 | 33 | 10
units on a scale | -2.43 (0.10) | -2.55 (0.19) | -1.66 (0.13) | -1.50 (0.25)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.577, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.567, Mixed Models Analysis — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 8:Retardation
Description: Measures slowness of thought and speech; impaired ability to concentrate; decreased motor activity on a scale of 0 (normal speech and thought) to 4 (complete stupor).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.72 (0.04) | -0.69 (0.07) | -0.66 (0.04) | -0.51 (0.07)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.89 (0.05) | -0.90 (0.09) | -1.66 (0.13) | -1.50 (0.25)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.670, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.059, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.930, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.567, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

12. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 9:Agitation
Description: Measures agitation on a scale of 0 (none) to 4 (hand-wringing, nail-biting)
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.47 (0.04) | -0.48 (0.07) | -0.44 (0.05) | -0.41 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.53 (0.07) | -0.61 (0.12) | -0.57 (0.11) | -0.78 (0.21)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.896, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.796, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.381, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

13. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 10:Anxiety (Psychic)
Description: Measures anxiety on a scale of 0 (no difficulty) to 4 (fears expressed)
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -1.15 (0.06) | -0.90 (0.10) | -1.15 (0.06) | -0.81 (0.10)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.23 (0.12) | -1.13 (0.20) | -1.41 (0.12) | -1.70 (0.22)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.665, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.253, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

14. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 11:Anxiety (Somatic)
Description: Measures physiological concomitants of anxiety on a scale of 0 (absent) to 4 (incapacitating).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.61 (0.05) | -0.65 (0.09) | -0.68 (0.06) | -0.57 (0.10)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.98 (0.11) | -0.94 (0.19) | -1.20 (0.08) | -1.18 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.312, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.853, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.913, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

15. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 12:Somatic Symptoms/Gastrointestinal
Description: Measures gastrointestical somatic symptoms on a scale of 0 (none) to 2 (difficulty eating, requires medication for symptoms).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.44 (0.03) | -0.52 (0.06) | -0.40 (0.03) | -0.32 (0.05)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.98 (0.11) | -0.94 (0.19) | -0.46 (0.05) | -0.47 (0.09)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.234, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.216, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.853, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.908, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

16. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 13:Somatic Symptoms/General
Description: Measures general somatic symptoms on a scale of 0 (none) to 2 (any clear-cut symptoms).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.91 (0.05) | -0.88 (0.09) | -0.75 (0.05) | -0.49 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.36 (0.11) | -1.18 (0.20) | -0.94 (0.13) | -0.83 (0.25)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.414, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.717, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

17. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 14:Genital Symptoms
Description: Measures genital symptoms (loss of libido, menstrual disturbances) on a scale of 0 (absent) to 2 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.57 (0.05) | -0.54 (0.09) | -0.55 (0.06) | -0.40 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.89 (0.13) | -0.77 (0.22) | -0.68 (0.08) | -0.30 (0.15)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.780, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.152, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.637, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

18. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 15:Hypochondriasis
Description: Measures hypochondriasis on a scale of 0 (not present) to 4 (hypochondriacal delusions).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.36 (0.04) | -0.41 (0.06) | -0.52 (0.05) | -0.41 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.44 (82.99) | -0.53 (144.40) | -0.61 (0.09) | -0.41 (0.16)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.517, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

19. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 16:Loss of Weight
Description: Measures weight loss since last visit on a scale of 0 (no weight loss) to 2 (definite weight loss caused by present illness).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.21 (0.02) | -0.20 (0.04) | -0.25 (0.02) | -0.24 (0.04)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.44 (82.99) | -0.53 (144.40) | -0.61 (0.09) | -0.41 (0.16)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.741, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.722, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

20. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 17:Insight
Description: Measures insight on a scale of 0 (acknowledges being depressed and ill) to 2 (denies being ill at all).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.08 (0.01) | -0.07 (0.02) | -0.01 (0.01) | -0.01 (0.02)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.44 (82.99) | -0.53 (144.40) | -0.61 (0.09) | -0.41 (0.16)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.949, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

21. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 18A:Diurnal Variation
Description: Measures whether symptoms are worse in morning or evening on a scale of 0 (no variation), 1 (worse in morning), or 2 (worse in evening).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.32 (0.05) | -0.36 (0.09) | -0.45 (0.05) | -0.13 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.56 (0.12) | -0.26 (0.20) | -0.77 (0.13) | -0.70 (0.25)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.682, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.200, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.813, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

22. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 18B:Diurnal Variation-Severity
Description: Measures the severity of the diurnal variation on a scale of 0 (none) to 2 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.43 (0.04) | -0.49 (0.07) | -0.42 (0.05) | -0.21 (0.08)
  9 Month Change (n=29, n=8, n=32, n=10) | -0.60 (0.07) | -0.54 (0.12) | -0.63 (0.08) | -0.56 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.438, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

23. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 19: Depersonalization and Derealization
Description: Measures feelings of unreality on a scale of 0 (absent) to 4 (incapacitating).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.19 (0.02) | -0.21 (0.03) | -0.15 (0.02) | -0.14 (0.03)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.60 (0.07) | -0.54 (0.12) | -0.63 (0.08) | -0.56 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.588, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.758, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

24. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 20:Paranoid Symptoms
Description: Measures paranoid symptoms on a scale of 0 (none) to 2 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.15 (0.02) | -0.12 (0.04) | -0.13 (0.02) | -0.11 (0.03)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.60 (0.07) | -0.54 (0.12) | -0.63 (0.08) | -0.56 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.507, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.466, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

25. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 21:Obsessional and Compulsive Symptoms
Description: Measures obsessional and compulsive symptoms on a scale of 0 (absent) to 2 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.08 (0.02) | -0.06 (0.03) | -0.04 (0.02) | -0.06 (0.03)
  9 Month Change (n=29, n=9, n=33, n=10) | -0.60 (0.07) | -0.54 (0.12) | -0.63 (0.08) | -0.56 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.487, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.678, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

26. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 22B:Helplessness
Description: Measures feelings of helplessness on a scale of 0 (absent) to 4 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.95 (0.05) | -0.88 (0.09) | -0.98 (0.06) | -0.81 (0.10)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.16 (0.09) | -0.90 (0.16) | -1.34 (9.63) | -1.24 (17.77)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.505, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.135, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

27. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 23B:Hopelessness
Description: Measures feelings of hopelessness on a scale of 0 (absent) to 4 (expresses feelings of discouragement, despair, and/or pessimism about the future which cannot be dispelled).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -0.87 (0.05) | -0.74 (0.08) | -0.80 (0.05) | -0.51 (0.08)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.23 (0.08) | -1.34 (0.15) | -0.92 (0.07) | -0.85 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.576, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.676, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

28. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in HAMD-24 - Item 24B:Worthlessness
Description: Measures feelings of worthlessness on a scale of 0 (absent) to 4 (severe).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -1.00 (0.06) | -0.95 (0.09) | -0.95 (0.06) | -0.79 (0.09)
  9 Month Change (n=29, n=9, n=33, n=10) | -1.23 (0.08) | -1.34 (0.15) | -0.92 (0.07) | -0.85 (0.14)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.675, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.576, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.676, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

29. Secondary Outcome: Change From Baseline to 12 Week Endpoint in 30-Item Brief Profile of Mood States (BPOMS) Scale and Subscales (Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment).
Description: The 30-item BPOMS measures mood states and has 6 factors: tension-anxiety, depression-dejection, anxiety-hostility, fatigue, confusion, and vigor. Item scores: 0 (not at all) to 4 (extremely). Each factor scores range from 0 to 20. The Total score is sum of all factor scores minus the factor score for vigor (Total=Ten+Dep+Ang+Fat+Con-Vig).
Time Frame: Baseline, 12 weeks
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 193 | 58 | 193 | 63
units on a scale
  Total Score (n=192,n=54,n=185,n=61) | -26.41 (1.44) | -18.88 (2.38) | -28.67 (1.52) | -22.67 (2.37)
  Tension-Anxiety (n=193,n=58,n=193,n=62) | -4.37 (0.26) | -3.20 (0.44) | -4.61 (0.30) | -4.05 (0.49)
  Depression-Dejection (n=193,n=58,n=191,n=62) | -6.30 (0.33) | -4.64 (0.55) | -6.78 (0.34) | -5.03 (0.53)
  Anger-Hostility (n=193,n=58,n=192,n=63) | -4.46 (0.28) | -3.09 (0.46) | -4.94 (0.30) | -3.63 (0.48)
  Vigor-Activity (n=192,n=55,192,n=63) | 2.55 (0.29) | 1.82 (0.49) | 2.57 (0.32) | 1.48 (0.51)
  Fatigue-Inertia (n=193,n=57,n=190,n=63) | -5.30 (0.36) | -4.68 (0.59) | -6.08 (0.37) | -5.54 (0.59)
  Confusion-Bewilderment (n=192,n=58,n=189,n=62) | -3.62 (0.23) | -2.86 (0.39) | -3.56 (0.25) | -3.10 (0.40)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Total Score (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Tension-Anxiety (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.324, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Depression-Dejection (Change=Endpoint minus baseline)
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Anger-Hostility (Change=Endpoint minus baseline)
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 7]
Statistical Analysis 9: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.201, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Vigor-Activity (Change=Endpoint minus baseline)
Statistical Analysis 10: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 9]
Statistical Analysis 11: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.368, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Fatigue-Inertia (Change=Endpoint minus baseline)
Statistical Analysis 12: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.435, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 11]
Statistical Analysis 13: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Confusion-Bewilderment (Change=Endpoint minus baseline)
Statistical Analysis 14: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.313, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 13]

30. Secondary Outcome: Change From Baseline to 9 Month Endpoint in 30-Item Brief Profile of Mood States (BPOMS) Scale and Subscales (Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment)
Description: as for outcome 29
Time Frame: Baseline, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 29 | 9 | 33 | 9
units on a scale
  Total Score | -25.67 (2.83) | -22.99 (4.89) | -28.39 (2.46) | -25.51 (4.68)
  Tension-Anxiety | -5.36 (0.51) | -4.18 (0.88) | -4.68 (0.50) | -3.50 (0.94)
  Depression-Dejection | -7.60 (0.60) | -6.49 (1.04) | -7.18 (0.63) | -5.56 (1.24)
  Anger-Hostility | -4.34 (0.60) | -3.38 (1.04) | -5.98 (0.40) | -4.99 (0.73)
  Vigor-Activity | 2.63 (0.78) | 3.11 (1.39) | 2.00 (0.74) | 3.04 (1.42)
  Fatigue-Inertia | -7.43 (0.73) | -7.40 (1.26) | -6.34 (0.59) | -7.03 (1.17)
  Confusion-Bewilderment | -3.95 (0.45) | -2.47 (0.79) | -3.54 (0.35) | -3.07 (0.64)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.639, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.584, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.251, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.265, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.366, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 5]
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.426, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 7]
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.234, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 7]
Statistical Analysis 9: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.765, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 9]
Statistical Analysis 10: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.522, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 9]
Statistical Analysis 11: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.986, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 11]
Statistical Analysis 12: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.602, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 11]
Statistical Analysis 13: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.110, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 13]
Statistical Analysis 14: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.505, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Confusion-Bewilderment(Change=Endpoint minus baseline)

31. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Sheehan Disability Scale (SDS) Total Score and Subscores
Description: The SDS is completed by the patient and is used to assess the effect of the patient's symptoms on their work/social/family life. Individual item scores range from 0 to 10. Total scores range from 0 to 30 with higher values indicating greater disruption in the patient's work/social/family life.
Time Frame: Baseline, 12 weeks
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  Work Life (n=133,n=43,n=140,n=49) | -2.47 (0.22) | -2.12 (0.34) | -1.98 (0.22) | -1.22 (0.36)
  Social Life (n=194,n=59,n=195,n=63) | -2.93 (0.19) | -2.50 (0.31) | -2.67 (0.19) | -1.97 (0.30)
  Family Life (n=194,n=59,n=195,n=63) | -2.81 (0.19) | -2.19 (0.32) | -2.66 (0.19) | -1.56 (0.31)
  Total Score (n=195,n=59,n=195,n=63) | -8.32 (0.53) | -6.84 (0.87) | -7.70 (0.52) | -4.94 (0.84)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.366, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Work Life (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.065, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.229, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Social Life (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.092, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Family Life (Change=Endpoint minus baseline)
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Total Score(Change=Endpoint minus baseline)
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]

32. Secondary Outcome: Change From Baseline to 9 Month Endpoint in Sheehan Disability Scale (SDS) Total Score and Subscores
Description: as for outcome 31
Time Frame: Baseline, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 29 | 9 | 33 | 10
units on a scale
  Work Life (n=22, n=8, n=22, n=7) | -3.88 (0.69) | -4.01 (1.10) | -2.26 (0.37) | -2.16 (0.66)
  Social Life (n=29, n=9, n=33, n=10) | -4.15 (0.37) | -4.35 (0.65) | -3.88 (0.33) | -3.66 (0.62)
  Family Life (n=29, n=9, n=33, n=10) | -3.46 (0.36) | -2.99 (0.64) | -3.30 (0.34) | -3.07 (0.66)
  Total Score (n=29, n=9, n=33, n=10) | -11.60 (1.02) | -11.15 (1.79) | -9.42 (0.97) | -8.67 (1.88)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.921, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.895, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.761, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.519, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 5]
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.755, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.829, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]

33. Secondary Outcome: Path Analysis of BPOMS Total Score to Overall Improvement in HAMD-24 Item 7
Description: Relative contribution of improvement on the mood states, defined by BPOMS total score (calculated from subscales) to overall improvement in work and activities, HAMD-24 item 7 using path analysis.
Time Frame: Over 12 weeks
Measure: Number; unit: coefficient
Groups:
- Group A - Ordinary Coefficient; Group B - Ordinary Coefficient: Mathematical estimate of the relationship between the dependent variable and the independent variable from linear regression in the Duloxetine 60 mg group.
- Group A - Standardized Coefficient; Group B - Standardized Coefficient: Mathematical estimate of the relationship between the dependent variable and the independent variable from linear regression expressed in units of standard deviation in the Duloxetine 60 mg group.
Arm/Group | Group A - Ordinary Coefficient | Group A - Standardized Coefficient | Group B - Ordinary Coefficient | Group B - Standardized Coefficient
Number analyzed (Participants) | 214 | 102 | 220 | 110
coefficient
  Direct Treatment Effect | -0.032 | -0.012 | 0.219 | 0.087
  Indirect Treatment Effect from BPOMS Total Score | 0.376 | 0.145 | 0.209 | 0.083
  Total Treatment Effect | 0.343 | 0.132 | 0.428 | 0.170
Statistical Analysis 1: Comparison: Group A - Ordinary Coefficient vs Group A - Standardized Coefficient; Test type: Superiority or Other; p = 0.753, Regression, Linear — P-value for Direct Treatment Effect
Statistical Analysis 2: Comparison: Group B - Ordinary Coefficient vs Group B - Standardized Coefficient; Test type: Superiority or Other; p = 0.036, Regression, Linear — P-value for Direct Treatment Effect

34. Secondary Outcome: Path Analysis of BPOMS Total Score to Overall Improvement in HAMD-24 Item 7 - Percent of Total Effect
Description: For Group A, at least one effect was in the opposite direction, percent of total effect was not calculated.
Time Frame: over 12 weeks
Measure: Number; unit: percent of total effect
Groups:
- Group B - Percent of Total Effect: The percentage of the total treatment effect explained by the direct and indirect effects of treatment in the duloxetine 60 mg group.
Arm/Group | Group B - Percent of Total Effect
Number analyzed (Participants) | 214
percent of total effect
  Direct Treatment Effect | 51.14
  Indirect Treatment Effect from BPOMS Total Score | 48.86
  Total Treatment Effect | 100.00

35. Secondary Outcome: Path Analysis of BPOMS Total Score to Overall Improvement in Sheehan Disability Scale (SDS) Total Score
Description: Relative contribution of improvement on the mood states, defined by BPOMS total score (determined from subscales) to overall improvement in SDS total score using path analysis.
Time Frame: over 12 weeks
Measure: Number; unit: coefficient
Arm/Group | Group A - Ordinary Coefficient | Group A - Standardized Coefficient | Group B - Ordinary Coefficient | Group B - Standardized Coefficient
Number analyzed (Participants) | 214 | 102 | 220 | 110
coefficient
  Direct Treatment Effect | -0.577 | -0.032 | 0.955 | 0.052
  Indirect Treatment Effect from BPOMS Total Score | 2.754 | 0.151 | 1.761 | 0.095
  Total Treatment Effect | 2.177 | 0.120 | 2.716 | 0.147
Statistical Analysis 1: Comparison: Group A - Ordinary Coefficient vs Group A - Standardized Coefficient; Test type: Superiority or Other; p = 0.342, Regression, Linear — P-value for Direct Treatment Effect
Statistical Analysis 2: Comparison: Group B - Ordinary Coefficient vs Group B - Standardized Coefficient; Test type: Superiority or Other; p = 0.111, Regression, Linear — P-value for Direct Treatment Effect

36. Secondary Outcome: Path Analysis of BPOMS Total Score to Overall Improvement in SDS Total Score - Percent of Total Effect
Description: For Group A, at least one effect was in the opposite direction, percent of total effect was not calculated.
Time Frame: Over 12 weeks
Measure: Number; unit: percent of total effect
Arm/Group | Group B - Percent of Total Effect
Number analyzed (Participants) | 214
percent of total effect
  Direct Treatment Effect | 35.17
  Indirect Treatment Effect from BPOMS Total Score | 64.83
  Total Treatment Effect | 100.00

37. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in 16-Item Quick Inventory of Depressive Symptomatology Self Report (QIDS16SR) Total Score
Description: A 16-item patient-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity.
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 58 | 194 | 62
units on a scale
  12 Week Change | -6.31 (0.34) | -5.65 (0.55) | -6.54 (0.33) | -5.21 (0.52)
  9 Month Change (n=29, n=9, n=33, n=9) | -8.41 (0.77) | -6.85 (1.36) | -7.17 (0.59) | -6.15 (1.11)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.302, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.325, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 3]

38. Secondary Outcome: Probability of Remission at 12 Week Endpoint and Sustained Remission at 9 Month Endpoint
Description: Probability of remission as measured by the HAMD17 Total Score ≤ 7 and by the QIDS16SR Total Score ≤ 5. The visitwise percentages of patients meeting criteria in the Acute Therapy Phase for remission (visitwise binary outcome, yes/no) will be analyzed using a categorical, pseudo-likelihood-based repeated measures approach. This analysis will include the fixed, categorical effects of treatment, investigator, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline score.
Time Frame: 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: probability of remission
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
probability of remission
  12 Week HAMD-17 Total (n=194,n=59,n=195,n=64) | 0.38 (0.21) | 0.35 (0.31) | 0.35 (0.19) | 0.18 (0.34)
  12 Week QIDS16 Total Score (n=194,n=58,n=194,n=62) | 0.30 (0.19) | 0.30 (0.30) | 0.33 (0.17) | 0.19 (0.30)
  9 Month HAMD-17 Total Score (n=29,n=9,n=33,n=10) | 0.63 (0.35) | 0.62 (0.63) | 0.70 (0.36) | 0.57 (0.65)
  9 Month QIDS16 Total Score (n=29,n=9,n=33,n=9) | 0.71 (0.31) | 0.54 (0.51) | 0.71 (0.35) | 0.64 (0.66)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.731, Mixed Models Analysis — P-value for 12 Week HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — P-value for 12 Week HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.948, Mixed Models Analysis — P-value for 12 Week QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — P-value for 12 Week QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis — P-value for 9 Month HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.442, Mixed Models Analysis — P-value for 9 Month HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.218, Mixed Models Analysis — P-value for 9 Month QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.648, Mixed Models Analysis — P-value for 9 Month QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit

39. Secondary Outcome: Probability of Response at 12 Week Endpoint
Description: Probability of response as measured by ≥ 50% Improvement in the HAMD17 Total Score and ≥ 50% Improvement in the QIDS16SR Total Score. The visitwise percentages of patients meeting criteria in the Acute Therapy Phase for response (visitwise binary outcome, yes/no) will be analyzed using a categorical, pseudo-likelihood-based repeated measures approach. This analysis will include the fixed, categorical effects of treatment, investigator, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline score.
Time Frame: 12 weeks
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: probability of response
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
probability of response
  HAMD-17 Total Score (n=194,n=59,n=195,n=64) | 0.63 (0.16) | 0.60 (0.27) | 0.63 (0.16) | 0.46 (0.26)
  QIDS16 Total Score (n=194,n=58,n=194,n=62) | 0.44 (0.15) | 0.41 (0.26) | 0.45 (0.16) | 0.34 (0.26)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.653, Mixed Models Analysis — P-value for 12 week HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — P-value for 12 week HAMD-17. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.665, Mixed Models Analysis — P-value for 12 week QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis — P-value for 12 week QIDS16. Model=Baseline, Pooled Investigator, Visit, Treatment, and Treatment*Visit

40. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in Pain Numerical Rating Scale (NRS)
Description: Item 1=Average musculoskeletal pain severity over the last week as measured by an 11-point Likert scale. Scores range from 0 (no pain) to 10 (worst possible pain). Item 7=How much they have been bothered by pain over the last week. Scores range from 0 (not bothered at all)to 10 (extremely bothered).
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 193 | 63
units on a scale
  Item 1 - 12 Week Change | -1.14 (0.16) | -1.35 (0.26) | -0.96 (0.18) | -1.16 (0.30)
  Item 7 - 12 Week Change | -1.33 (0.17) | -1.73 (0.27) | -1.14 (0.18) | -1.36 (0.30)
  Item 1 - 9 Month Change (n=29, n=9, n=33, n=10) | -1.30 (0.41) | -0.10 (0.73) | -2.10 (0.41) | -2.36 (0.75)
  Item 7 - 9 Month Change (n=29, n=9, n=33, n=10) | -1.56 (0.42) | -0.42 (0.74) | -2.24 (0.35) | -2.11 (0.64)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.475, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Item 1 Average Pain Severity 12 Week Change (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.561, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.213, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Item 7 How Bothered by Pain 12 Week Change (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.536, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Item 1 Average Pain Severity 9 Month Change (Change=Endpoint minus baseline)
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.759, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.190, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Item 7 How Bothered by Pain 9 Month Change (Change=Endpoint minus baseline)
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.852, Mixed Models Analysis — [p-value comment as in outcome 40, analysis 7]

41. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoint in the Clinical Global Impression-Severity Scale (CGI-S)
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 195 | 64
units on a scale
  12 Week Change | -1.93 (0.08) | -1.58 (0.14) | -1.97 (0.09) | -1.25 (0.15)
  9 Month Change (n=29, n=9, n=33, n=10) | -2.14 (0.22) | -1.97 (0.40) | -2.61 (0.21) | -2.23 (0.37)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.705, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.388, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

42. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH-CPFQ)
Description: A 7-item patitent-rated questionnaire pertaining to a patient's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each of the 7 questions is scored on a 6-point scale ranging fom 1 (greater than normal) to 6 (totally absent). Total score ranges from 7 to 42.
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 193 | 59 | 194 | 64
units on a scale
  12 Week Change | -7.60 (0.46) | -6.39 (0.74) | -7.96 (0.47) | -6.85 (0.74)
  9 Month Change (n=29, n=9, n=32, n=10) | -7.17 (0.88) | -7.13 (1.54) | -8.19 (0.84) | -6.77 (1.48)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.198, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.982, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.407, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

43. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in the Social Adaptation Self-evaluation Scale (SASS) Total Score
Description: A 21-item self-rated scale that evaluates patient social motivation and behavior in depression. Each of the 21 items is scored from 0 (minimal social adjustment) to 3 (maximal social adjustment). Total score ranges from 0 to 60.
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 187 | 57 | 185 | 62
units on a scale
  12 Week Change | 7.18 (0.62) | 3.40 (0.99) | 7.54 (0.61) | 4.52 (0.92)
  9 Month Change (n=28, n=9, n=30, n=10) | 8.00 (1.14) | 5.30 (1.92) | 13.81 (1.04) | 9.28 (1.92)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.231, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

44. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in Blood Pressure
Description: Sitting systolic and diastolic blood pressure.
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 58 | 196 | 63
mm Hg
  Systolic Blood Pressure (SBP) - 12 Week Change | -0.12 (0.78) | 0.05 (1.33) | 0.73 (0.76) | -2.95 (1.25)
  Diastolic Blood Pressure (DBP) - 12 Week Change | 0.48 (0.51) | -0.58 (0.88) | 1.97 (0.61) | -0.50 (1.00)
  SBP - 9 Month Change (n=28, n=9, n=33, n=10) | -1.18 (2.31) | -0.44 (4.02) | -2.22 (1.63) | -0.54 (2.91)
  DBP - 9 Month Change (n=28, n=9, n=33, n=10) | -2.25 (1.25) | 1.46 (2.18) | -1.52 (1.47) | -1.05 (2.69)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.914, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Systolic Blood Pressure 12 Week Change (Change=Endpoint minus baseline)
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.296, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Diastolic Blood Pressure 12 Week Change (Change=Endpoint minus baseline)
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 3]
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.874, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Systolic Blood Pressure (SBP) 9 Month Change (Change=Endpoint minus baseline)
Statistical Analysis 6: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.614, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 5]
Statistical Analysis 7: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.146, Mixed Models Analysis — Model: Change from baseline=Baseline, Pooled Investigator, Visit, Treatment, Treatment*Visit and Baseline*Visit. P-value for Diastolic Blood Pressure (DBP) 9 Month Change (Change=Endpoint minus baseline)
Statistical Analysis 8: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.877, Mixed Models Analysis — [p-value comment as in outcome 44, analysis 7]

45. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in Pulse Rate
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 58 | 196 | 63
beats per minute
  12 Week Change | 1.40 (0.57) | -1.52 (1.01) | 0.68 (0.70) | -2.05 (1.18)
  9 Month Change (n=28, n=9, n=33, n=10) | 1.08 (1.79) | -0.30 (3.11) | 1.18 (1.17) | -3.04 (2.05)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.701, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

46. Secondary Outcome: Change From Baseline to 12 Week and 9 Month Endpoints in Weight
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 58 | 195 | 63
kilograms
  12 Week Change | -0.54 (0.20) | 0.38 (0.31) | -0.38 (0.20) | -0.23 (0.30)
  9 Month Change (n=28, n=9, n=33, n=10) | -1.18 (2.31) | -0.44 (4.02) | -0.94 (0.55) | 0.06 (1.02)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.672, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.874, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 3]

47. Secondary Outcome: Abnormal Vital Signs at Anytime Over 12 Weeks
Time Frame: over 12 weeks
Population: Number of participants wtih a normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 250 | 120 | 254 | 128
participants
  Sitting Pulse Rate - High | 1 | 0 | 1 | 0
  Weight - Gain | 0 | 0 | 0 | 0
  Weight - Loss | 0 | 1 | 2 | 0
  Sitting Systolic Blood Pressure - High | 3 | 1 | 6 | 0
  Sitting Diastolic Blood Pressure - High | 2 | 0 | 2 | 3

48. Secondary Outcome: Abnormal Vital Signs at Anytime Over 9 Months
Time Frame: over 9 months
Population: Number of participants with a normal baseline and at least oone post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 250 | 120 | 254 | 128
participants
  Sitting Pulse - High | 1 | 0 | 2 | 0
  Weight - Gain | 2 | 0 | 3 | 0
  Weight - Loss | 5 | 1 | 5 | 0
  Sitting Systolic Blood Pressure - High | 4 | 2 | 7 | 0
  Sitting Diastolic Blood Pressure - High | 2 | 0 | 4 | 3

49. Secondary Outcome: Abnormal Vital Signs at 12 Week Endpoint
Time Frame: 12 weeks
Population: Number of participants with a normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 250 | 120 | 254 | 128
participants
  Sitting Pulse Rate - High | 0 | 0 | 1 | 0
  Weight - Gain | 0 | 0 | 0 | 0
  Weight - Loss | 0 | 1 | 2 | 0
  Sitting Systolic Blood Pressure - High | 0 | 0 | 4 | 0
  Sitting Diastolic Blood Pressure - High | 0 | 0 | 0 | 1

50. Secondary Outcome: Abnormal Vital Signs at 9 Month Endpoint
Time Frame: 9 months
Population: Number of participants with a normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 250 | 120 | 254 | 128
participants
  Sitting Pulse - High | 0 | 0 | 1 | 0
  Weight - Gain | 2 | 0 | 3 | 0
  Weight - Loss | 5 | 1 | 4 | 0
  Sitting Systolic Blood Pressure - High | 1 | 0 | 4 | 0
  Sitting Diastolic Blood Pressure - High | 0 | 0 | 0 | 1

51. Secondary Outcome: Statistically Significant Changes in Baseline to 12 Week and 9 Month Endpoints Laboratory Values - Bilirubin, Creatinine, Uric Acid
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and at least one post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: micromole per Liter
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 214 | 102 | 220 | 110
micromole per Liter
  Bilirubin - 12 Week Change | 0.10 (4.09) | -0.19 (3.63) | -0.51 (3.92) | 0.13 (3.64)
  Creatinine - 12 Week Change | -1.56 (9.55) | -0.85 (8.27) | -1.21 (8.95) | 0.82 (7.85)
  Uric Acid - 12 Week Change | -2.77 (48.20) | 5.74 (41.92) | -12.36 (46.02) | 7.05 (44.20)
  Bilirubin - 9 Month Change (n=193,n=60,n=202,n=66) | -0.13 (4.04) | -0.12 (2.94) | -0.56 (3.77) | 0.25 (3.56)
  Uric Acid - 9 Month Change (n=193,n=60,n=202,n=66) | -2.11 (48.77) | -2.25 (42.59) | -8.66 (47.85) | 6.50 (44.80)
Statistical Analysis 1: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.046, ANOVA — P-value for Bilirubin - 12 Week Change
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.031, ANOVA — P-value for Creatinine - 12 Week Change
Statistical Analysis 3: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.003, ANOVA — P-value for Uric Acid - 12 Week Change
Statistical Analysis 4: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.033, ANOVA — P-value for Bilirubin - 9 Month Change
Statistical Analysis 5: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.013, ANOVA — P-value for Uric Acid - 9 Month Change

52. Secondary Outcome: Statistically Significant Changes in Baseline to 12 Week and 9 Month Endpoints Laboratory Values - Hematocrit
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and at least one post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: Proportion of 1.0
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 191 | 57 | 196 | 67
Proportion of 1.0
  Hematocrit - 12 Week Change | -0.00 (0.03) | -0.01 (0.03) | 0.00 (0.03) | -0.01 (0.03)
  Hematocrit - 9 Month Change (n=194,n=59,=197,n=67) | -0.00 (0.03) | -0.00 (0.03) | 0.00 (0.03) | -0.01 (0.03)
Statistical Analysis 1: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.037, ANOVA — P-value for Hematocrit - 12 Week Change
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.029, ANOVA — P-value for Hematocrit - 9 Month Change

53. Secondary Outcome: Statistically Significant Changes in Baseline to 12 Week and 9 Month Endpoints Laboratory Values - Mean Cell Volume (MCV)
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and at least one post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: femtoliter
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 191 | 57 | 196 | 67
femtoliter
  MCV - 12 Week Change | 0.98 (2.85) | 1.30 (3.30) | 0.71 (3.23) | -0.47 (3.18)
  MCV - 9 Month Change (n=194,n=59,n=197,n=67) | 1.07 (2.90) | 1.66 (3.08) | 0.88 (3.36) | -0.31 (3.48)
Statistical Analysis 1: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.013, ANOVA — P-value for MCV - 12 Week Change
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.014, ANOVA — P-value for MCV - 9 Month Change

54. Secondary Outcome: Statistically Significant Changes in Baseline to 12 Week and 9 Month Endpoints Laboratory Values - Chloride, Urea Nitrogen, Cholesterol, Sodium
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and at least one post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: millimole per Liter
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 192 | 58 | 202 | 66
millimole per Liter
  Chloride - 12 Week Change | -0.80 (2.85) | 0.24 (2.62) | -0.91 (2.75) | -0.39 (2.51)
  Urea Nitrogen - 12 Week Change | -0.06 (1.29) | 0.26 (1.04) | 0.01 (1.20) | 0.15 (1.38)
  Chloride - 9 Month Change (n=193,n=60,n=202,n=66) | -0.74 (2.92) | 0.54 (2.44) | -0.82 (2.71) | -0.31 (2.40)
  Cholesterol - 9 Month (n=193,n=60,n=202,n=66) | -0.06 (0.70) | -0.30 (0.78) | 0.04 (0.75) | -0.08 (0.51)
  Sodium - 9 Month Change (n=193,n=60,n=202,n=66) | -1.67 (3.30) | -0.73 (2.47) | -1.86 (3.16) | -1.73 (3.12)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.022, ANOVA — P-value for Chloride - 12 Week Change
Statistical Analysis 2: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.044, ANOVA — P-value for Urea Nitrogen - 12 Week Change
Statistical Analysis 3: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.004, ANOVA — P-value for Chloride - 9 Month Change
Statistical Analysis 4: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.045, ANOVA — P-value for Cholesterol - 9 Month Change
Statistical Analysis 5: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.043, ANOVA — P-value for Sodium - 9 Month Change

55. Secondary Outcome: Statistically Significant Changes in Baseline to 12 Week and 9 Month Endpoints Laboratory Values - Platelet Count
Time Frame: Baseline, 12 weeks, 9 months
Population: Number of participants with non-missing data at baseline and at least post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: Billions per Liter
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 187 | 56 | 193 | 67
Billions per Liter
  12 Week Change | 8.11 (37.00) | -7.10 (38.83) | 10.55 (37.53) | 12.02 (51.41)
  9 Month Change (n=191, n=58, n=194, n=67) | 8.06 (37.62) | -10.17 (35.73) | 5.96 (39.44) | 10.18 (51.19)
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.017, ANOVA — P-value for 12 Week Change
Statistical Analysis 2: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.003, ANOVA — P-value for 9 Month Change

56. Secondary Outcome: Statistically Significant Changes in Baseline to 9 Month Endpoint Laboratory Values - Alkaline Phosphatase
Time Frame: baseline, 9 months
Population: Number of participants with non-missing data at baseline and at least one post baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 193 | 60 | 202 | 66
Units per Liter | -0.18 (10.61) | -2.30 (10.20) | 0.23 (10.94) | -3.75 (8.19)
Statistical Analysis 1: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.033, ANOVA

57. Secondary Outcome: Statistically Significant Changes in Baseline to 9 Month Endpoint Laboratory Values - Hemoglobin
Time Frame: Baseline, 9 months
Population: Number of participants with non-missing data at baseline and at least one post-baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: millimoles per Liter (iron)
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 197 | 67
millimoles per Liter (iron) | -0.13 (0.45) | -0.19 (0.54) | -0.01 (0.47) | -0.17 (0.53)
Statistical Analysis 1: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.045, ANOVA

58. Secondary Outcome: Statistically Significant Abnormal Laboratory Values at Anytime/12 Week Endpoint
Description: The number of participants with statistically significant abnormal lab values at anytime and at 12 week endpoint were the same.
Time Frame: over 3 months
Population: Number of participants with a normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 191 | 57 | 201 | 66
participants
  Lymphocytes - High (n=186,n=57,n=195,n=66) | 1 | 3 | 2 | 1
  Potassium - Low (n=191,n=57,n=201,n=66) | 0 | 0 | 1 | 3
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.041, Fisher Exact — P-value for Lymphocytes - High
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.048, Fisher Exact — P-value for Potassium - Low

59. Secondary Outcome: Statistically Significant Abnormal Laboratory Values at Anytime During 9 Months
Time Frame: over 9 months
Population: Number of participants with a normal baseline at at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 194 | 59 | 202 | 67
participants
  Lymphocytes - High (n=189,n=59,n=196,n=66) | 1 | 4 | 2 | 1
  Potassium - Low (n=194,n=59,n=202,n=67) | 0 | 0 | 1 | 3
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.012, Fisher Exact — P-value for Lymphocytes - High
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.049, Fisher Exact — P-value for Potassium - Low

60. Secondary Outcome: Statistically Significant Abnormal Laboratory Values at 9 Month Endpoint
Time Frame: 9 months
Population: Number of participants with a normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Group A - Duloxetine | Group A - Placebo | Group B - Duloxetine | Group B - Placebo
Number analyzed (Participants) | 189 | 59 | 196 | 66
participants
  Lymphocytes - High (n=189,n=59,n=196,n=66) | 1 | 4 | 1 | 1
  Hemoglobin - Low (n=184,n=54,n=184,n=63) | 5 | 2 | 2 | 4
Statistical Analysis 1: Comparison: Group A - Duloxetine vs Group A - Placebo; Test type: Superiority or Other; p = 0.012, Fisher Exact — P-value for Lymphocytes - High
Statistical Analysis 2: Comparison: Group B - Duloxetine vs Group B - Placebo; Test type: Superiority or Other; p = 0.038, Fisher Exact — P-value for Hemoglobin - Low

61. Secondary Outcome: Summary of Adverse Events Leading to Discontinuation
Time Frame: over 9 months
Population: Number of randomized participants in each treatment group.
Measure: Number; unit: participants
Groups:
- Duloxetine (Not Escalated): duloxetine 60 mg every day (QD), by mouth (PO) for 3 months, after which participants remained on duloxetine 60 mg QD, PO for 6 months.
- Duloxetine (Escalated): duloxetine 60 mg every day (QD), by mouth (PO) for 3 months, after which participants were increased to duloxetine 120 mg QD, PO for 6 months
- Placebo (Not Rescued); Placebo (Rescued): placebo every day (QD), by mouth (PO) for up to 9 months, may be increased to duloxetine 60 mg QD, PO during the first 3 months as part of a rescue plan with pre-defined criteria (Patients meeting criteria will automatically be assigned to duloxetine 60 mg QD).
Arm/Group | Duloxetine (Not Escalated) | Duloxetine (Escalated) | Placebo (Not Rescued) | Placebo (Rescued)
Number analyzed (Participants) | 247 | 271 | 104 | 154
participants
  Nausea | 5 | 0 | 0 | 1
  Dizziness | 2 | 1 | 1 | 1
  Headache | 1 | 0 | 2 | 1
  Rash | 2 | 0 | 1 | 0
  Fatigue | 2 | 2 | 0 | 0
  Insomnia | 2 | 1 | 0 | 0
  Suicide attempt | 1 | 1 | 1 | 0
  Weight increased | 0 | 0 | 2 | 0
  Abdominal pain lower | 0 | 0 | 1 | 0
  Abnormal dreams | 1 | 0 | 0 | 0
  Asthma | 0 | 0 | 1 | 0
  Blood pressure increased | 1 | 0 | 0 | 0
  Chest pain | 1 | 0 | 0 | 0
  Completed suicide | 0 | 0 | 1 | 0
  Constipation | 2 | 1 | 0 | 0
  Crying | 0 | 0 | 1 | 0
  Depression | 0 | 1 | 1 | 0
  Diarrhoea | 1 | 1 | 0 | 1
  Disturbance in attention | 1 | 0 | 0 | 0
  Dry mouth | 1 | 0 | 0 | 0
  Dysgeusia | 1 | 0 | 0 | 0
  Hepatic function abnormal | 1 | 0 | 0 | 0
  Hernia | 1 | 0 | 0 | 0
  Hyperhidrosis | 1 | 0 | 0 | 0
  Hypertension | 1 | 1 | 0 | 1
  Influenza | 0 | 0 | 1 | 0
  Irritability | 1 | 0 | 1 | 0
  Lower gastrointestinal haemorrhage | 1 | 0 | 0 | 0
  Lower limb fracture | 0 | 0 | 1 | 0
  Mania | 1 | 0 | 0 | 0
  Migraine | 1 | 0 | 0 | 0
  Muscular weakness | 1 | 0 | 0 | 0
  Non-cardiac chest pain | 1 | 0 | 0 | 0
  Paranoia | 0 | 0 | 1 | 0
  Pregnancy | 1 | 0 | 0 | 0
  Restlessness | 1 | 0 | 0 | 0
  Road traffic accident | 1 | 0 | 0 | 0
  Ruptured cerebral aneurysm | 1 | 0 | 0 | 0
  Pneumonia | 1 | 0 | 0 | 1
  Tremor | 1 | 0 | 0 | 0
  Urinary hesitation | 0 | 0 | 1 | 0
  Urinary retention | 1 | 0 | 0 | 0
  Wound infection staphylococcal | 0 | 0 | 1 | 0
  Anorgasmia | 0 | 0 | 0 | 1
  Astigmatism | 0 | 1 | 0 | 0
  Cardiac failure congestive | 0 | 1 | 0 | 0
  Depressive symptom | 0 | 1 | 0 | 0
  Dyspepsia | 0 | 1 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0
  Hepatic enzyme increased | 0 | 1 | 0 | 0
  Libido decreased | 0 | 0 | 0 | 1
  Night sweats | 0 | 1 | 0 | 0
  Myocardial infarction | 0 | 0 | 0 | 1
  Nightmare | 0 | 1 | 0 | 0
  Palpitations | 0 | 0 | 0 | 1
  Pruritus | 0 | 0 | 0 | 1
  Sexual dysfunction | 0 | 1 | 0 | 0
  Somnolence | 1 | 0 | 0 | 0
  Sedation | 0 | 0 | 0 | 1
  Vomiting | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Groups:
- Duloxetine: duloxetine 60 mg every day (QD), by mouth (PO) for 3 months, after which may be increased to duloxetine 120 mg QD, PO for 6 months
- Placebo: placebo every day (QD), by mouth (PO) for up to 9 months, may be increased to duloxetine 60 mg QD, PO during the first 3 months as part of a rescue plan with pre-defined criteria (Patients meeting criteria will automatically be assigned to duloxetine 60 mg QD).
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 18 | 14
Other Adverse Events (participants affected / at risk) | 497 | 237
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine | Placebo
Cardiac failure congestive (Cardiac disorders) | 1/518 (1) | 0/258 (0)
Myocardial infarction (Cardiac disorders) | 0/518 (0) | 1/258 (1)
Pericardial effusion (Cardiac disorders) | 1/518 (1) | 0/258 (0)
Pericarditis (Cardiac disorders) | 1/518 (1) | 0/258 (0)
Colitis (Gastrointestinal disorders) | 1/518 (1) | 0/258 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/518 (0) | 1/258 (1)
Fatigue (General disorders) | 1/518 (1) | 0/258 (0)
Non-cardiac chest pain (General disorders) | 1/518 (1) | 0/258 (0)
Biliary colic (Hepatobiliary disorders) | 0/518 (0) | 1/258 (1)
Diverticulitis (Infections and infestations) | 0/518 (0) | 1/258 (1)
Gangrene (Infections and infestations) | 0/518 (0) | 1/258 (1)
Gastroenteritis (Infections and infestations) | 1/518 (1) | 0/258 (0)
Oesophageal candidiasis (Infections and infestations) | 0/518 (0) | 1/258 (1)
Pneumonia (Infections and infestations) | 1/518 (1) | 1/258 (1)
Pyelonephritis (Infections and infestations) | 1/518 (1) | 0/258 (0)
Sepsis (Infections and infestations) | 0/518 (0) | 1/258 (1)
Sinusitis (Infections and infestations) | 1/518 (1) | 0/258 (0)
Staphylococcal infection (Infections and infestations) | 1/518 (1) | 1/258 (1)
Subcutaneous abscess (Infections and infestations) | 1/518 (1) | 0/258 (0)
Tooth infection (Infections and infestations) | 1/518 (1) | 0/258 (0)
Urinary tract infection (Infections and infestations) | 0/518 (0) | 1/258 (1)
Wound infection staphylococcal (Infections and infestations) | 0/518 (0) | 1/258 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0/518 (0) | 1/258 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1/518 (1) | 0/258 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0/518 (0) | 1/258 (1)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/518 (1) | 0/258 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1/518 (1) | 0/258 (0)
Status migrainosus (Nervous system disorders) | 1/518 (1) | 0/258 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/518 (1) | 0/258 (0)
Completed suicide (Psychiatric disorders) | 0/518 (0) | 1/258 (1)
Depression (Psychiatric disorders) | 1/518 (1) | 1/258 (1)
Homicidal ideation (Psychiatric disorders) | 1/518 (1) | 0/258 (0)
Suicide attempt (Psychiatric disorders) | 2/518 (2) | 1/258 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1/518 (1) | 0/258 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/518 (0) | 1/258 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/518 (1) | 0/258 (0)
Deep vein thrombosis (Vascular disorders) | 1/518 (1) | 0/258 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine | Placebo
Hypothyroidism (Endocrine disorders) | 19/518 (19) | 15/258 (15)
Constipation (Gastrointestinal disorders) | 63/518 (71) | 30/258 (32)
Diarrhoea (Gastrointestinal disorders) | 62/518 (69) | 30/258 (33)
Dry mouth (Gastrointestinal disorders) | 95/518 (98) | 36/258 (38)
Dyspepsia (Gastrointestinal disorders) | 33/518 (34) | 16/258 (16)
Flatulence (Gastrointestinal disorders) | 24/518 (24) | 13/258 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 49/518 (49) | 26/258 (26)
Nausea (Gastrointestinal disorders) | 123/518 (155) | 37/258 (45)
Fatigue (General disorders) | 49/518 (52) | 20/258 (24)
Irritability (General disorders) | 22/518 (22) | 16/258 (17)
Seasonal allergy (Immune system disorders) | 65/518 (65) | 35/258 (35)
Nasopharyngitis (Infections and infestations) | 47/518 (48) | 19/258 (24)
Sinusitis (Infections and infestations) | 23/518 (24) | 18/258 (19)
Upper respiratory tract infection (Infections and infestations) | 38/518 (42) | 20/258 (25)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 44/518 (44) | 20/258 (20)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 8/518 (8) | 13/258 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39/518 (42) | 20/258 (21)
Arthritis (Musculoskeletal and connective tissue disorders) | 28/518 (28) | 9/258 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 79/518 (85) | 35/258 (36)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 28/518 (29) | 6/258 (6)
Dizziness (Nervous system disorders) | 58/518 (68) | 28/258 (30)
Headache (Nervous system disorders) | 177/518 (221) | 83/258 (96)
Migraine (Nervous system disorders) | 48/518 (51) | 18/258 (18)
Somnolence (Nervous system disorders) | 24/518 (25) | 13/258 (14)
Tension headache (Nervous system disorders) | 22/518 (25) | 14/258 (14)
Anxiety (Psychiatric disorders) | 27/518 (30) | 24/258 (28)
Insomnia (Psychiatric disorders) | 69/518 (72) | 38/258 (42)
Asthma (Respiratory, thoracic and mediastinal disorders) | 42/518 (43) | 19/258 (19)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 27/518 (27) | 6/258 (6)
Hypertension (Vascular disorders) | 100/518 (101) | 56/258 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days